CLINICAL TRIAL: NCT01316211
Title: Comparative Evaluation of Clinical Outcome in the Treatment of Degenerative Spinal Stenosis With Concomitant Low Back Pain by Decompression With and Without Additional Stabilization Using the Coflex™ Interlaminar Technology
Brief Title: Clinical Trial Comparing Decompression With and Without Coflex™ Interlaminar Technology Treating Lumbar Spinal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paradigm Spine (Industry)
Collaborators: MDT Medical Device Testing GmbH (Industry); MCRA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06k004
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Results first posted 2020-06-02 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Spinal Stenosis
Keywords: Back Pains; Pain, Back; Pains, Back; Backache; Backaches; Back Ache; Ache, Back; Aches, Back; Back Aches; Back Pain without Radiation; Vertebrogenic Pain Syndrome; Pain Syndrome, Vertebrogenic; Pain Syndromes, Vertebrogenic; Syndrome, Vertebrogenic Pain; Syndromes, Vertebrogenic Pain; Vertebrogenic Pain Syndromes; Back Pain with Radiation; Stenosis, spinal; Caudal stenosis; Spondylopathy; Spondylopathies; Low back pain; Lower back pain
MeSH Terms: conditions — Spinal Stenosis; Back Pain; Spinal Diseases; Low Back Pain | interventions — Decompression, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- coflex™ (Active Comparator): Implantation of coflex™ device in assigned patients
  Interventions: Device: Implantation of coflex™ after surgical decompression
- Surgical decompression (Active Comparator): Surgical decompression in patients with spinal stenosis without stabilization by an additional implant.
  Interventions: Procedure: Surgical decompression

INTERVENTIONS:
Device: Implantation of coflex™ after surgical decompression — The device will be implanted after surgical decompression in patients with spinal stenosis.
  Arms: coflex™
Procedure: Surgical decompression — Surgical decompression in patients with spinal stenosis without stabilization by an additional implant
  Arms: Surgical decompression

SUMMARY:
A 2 year comparative evaluation of clinical outcome in the treatment of degenerative spinal stenosis with concomitant low back pain by decompression with and without additional stabilization using the coflex® Interlaminar Technology

DETAILED DESCRIPTION:
The coflex® implant for interlaminar stabilization has been in clinical use for more than 10 years and is CE-certified according to the standards and approved in the United States.

This was a randomized multicenter study to collect prospective data for potential improvement in the therapy of low back pain during the treatment of spinal stenosis. The study was conducted in Germany.

ELIGIBILITY:
Inclusion Criteria:

1. Radiographic confirmation of clinical symptoms of at least moderate degenerative spinal stenosis, with constriction of the central spinal canal of one or two adjacent segments in the region L3 to L5 with the need for decompression.

   If necessary additional decompression in the adjacent segment(s) may be performed avoiding any instability in the affected segment.

   In addition the following may exist (but is not obligatory):
   * hypertrophy of the facet joints and subarticular recessus stenosis in the relevant segment or
   * stenosis of the foramen in the relevant segment
   * and/or stable retrolisthesis up to grade I verified by flexion-/extension X-ray films.
2. Radiographic confirmation of no translatory instability in the main segment as well as in adjacent segments (dynamic translatory instability ≤ 3 mm).
3. VAS back pain score of at least 50 mm on a 100 mm scale (for acute back pain or a period of at least 3 month of back pain before the onset of leg pain).
4. Minimum of 3 months conservative therapy without improvement of symptoms.
5. Age >40 years.
6. Oswestry Low Back Pain Disability Questionnaire score of at least 18/45 (40%) for German sites or 20/50 (40%) for the US sites (The question about sexual life will be excluded).
7. Suitability of the patient for a posterior surgery procedure.
8. Mental and physical ability of patient to follow the protocol according to compliance to time schedule, treatment plan, fill in of CRF pages and further study procedures.
9. Personally signed informed consent form before the start of any study related procedures.

Exclusion Criteria

Any of the following will exclude a subject from the study:

1. Preceding fusion or decompression surgery of the lumbar spine or preceding nucleotomy of the segments of concern (also if nucleotomy becomes necessary during surgery).
2. Radiographically confirmed damage of the vertebral body in the segment of concern in the lumbar spine (e.g. osteoporotic compression fracture or because of tumors)
3. Isthmic and degenerative spondylolisthesis (anterolisthesis; retrolisthesis > grade I) or spondylolysis (Pars fracture).
4. Degenerative lumbar scoliosis (> 25°).
5. Adipositas (obesity). Defined as a body mass index >40.
6. Pregnancy, or wish to get pregnant during the course of the study.
7. Known allergy for titanium and titanium alloys.
8. Fluoride infections - both systemic and local.
9. History of severe peripheral neuropathy.
10. Significant peripheral vascular disease (claudication intermittens ≥ stage 2b).
11. M. Paget or osteomalacia or other metabolic bone disorders.
12. Cauda equina syndrome.
13. Communicating diseases, including HIV, active hepatitis
14. Patients who are lawfully kept in an institution.
15. Subjects who, in the opinion of the investigator, will be inappropriate for inclusion into this clinical trial or will not comply with requirements of the study.
16. Subjects who participated in a clinical observation or therapy with X-ray during the last 10 years.
17. Subjects who participate(d) in another clinical trial (within the last 4 weeks) that might influence the safety and effectiveness assessment of this trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Germany (8):
  - Oberlinklinik Potsdam Orthopädische Fachklinik, Potsdam, Brandenburg
  - Orthopädische Universitätsklinik Frankfurt a.M., Frankfurt a.M., Hesse
  - Chirurgische Universitätsklinik Rostock Neurochirurgie, Rostock, Mecklenburg-Vorpommern
  - Otto-von-Guericke-Universität Magdeburg Klinik für Orthopädie, Magdeburg, Saxony-Anhalt
  - Ostseeklinik Damp Neurochirurgie, Damp, Schleswig-Holstein
  - Klinik für Neurochirurgie Lübeck, Lübeck, Schleswig-Holstein
  - Klinik für Wirbelsäulenchirurgie mit Skoliosezentrum Klinikum Neustadt, Neustadt, Schleswig-Holstein
  - Klinikum Ingolstadt Neurochirurgie, Ingolstadt

REFERENCES:
- [Derived] Schmidt S, Franke J, Rauschmann M, Adelt D, Bonsanto MM, Sola S. Prospective, randomized, multicenter study with 2-year follow-up to compare the performance of decompression with and without interlaminar stabilization. J Neurosurg Spine. 2018 Apr;28(4):406-415. doi: 10.3171/2017.11.SPINE17643. Epub 2018 Jan 26. PMID 29372860

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 120 patients in the Coflex group and 126 in the control group underwent surgery. 4 Coflex patients and 3 Control patients had to be excluded from full-analysis population, since no follow-up values were recorded and the reason of drop-out did not indicate treatment failure.
Period: Overall Study
Arm/Group | Coflex™ | Surgical Decompression
Started | 116 | 123
Completed | 105 | 111
Not Completed | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coflex™ | Surgical Decompression | Total
Number analyzed (Participants) | 116 | 123 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (9) | 68 (8) | 68 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 61 | 126
  Male | 51 | 62 | 113
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 116 | 123 | 239
Weight [Mean (Standard Deviation); unit: kg] | 84 (15) | 84 (17) | 84 (16.1)
Height [Mean (Standard Deviation); unit: cm] | 170 (9) | 170 (9) | 170 (9.4)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.0 (4.3) | 29.1 (4.7) | 29 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in ODI From Baseline to 24 Months
Description: The ODI, also known as the Oswestry Low Back Pain Disability Questionnaire is a questionnaire providing information on back and leg pain and the affects on managing everyday life by dividing questions into 10 sections. For this study, the questions on sexual activity will not be asked. The total possible score for each section is 0-5. The scores are then converted percentages ranging from 0% (minimal disability) to 100% (maximum possible disability).
Time Frame: Baseline, 3, 12, and 24 months
Measure: Mean (Standard Deviation); unit: percentage points
Arm/Group | Coflex™ | Surgical Decompression
Number analyzed (Participants) | 105 | 111
percentage points | -19.0 (2.1) | -22.5 (2.2)

2. Secondary Outcome: Number of Participants With Significant Migration or Expulsion of the Implant
Description: Assess significant migration, defined as > 5mm by x-ray images (point of reference is the tip of the U-portion implant identified on the corresponding x-ray image).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Coflex™
Number analyzed (Participants) | 105
Participants | 2

3. Secondary Outcome: Change in Visual Analog Scale (VAS) Back Pain From Baseline to 24 Months
Description: Improvement of the Visual Analog Scale (VAS) for low back pain (on the 100mm scale) compared to control group. 0 = no pain and 100 = worst pain imaginable.
Time Frame: Baseline, 3, 12, and 24 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Coflex™ | Surgical Decompression
Number analyzed (Participants) | 105 | 111
mm | -23.5 (2.8) | -23.1 (2.7)

4. Secondary Outcome: Change in Visual Analog Scale (VAS) Leg Pain From Baseline to 24 Months
Description: Improvement of the Visual Analog Scale (VAS) for leg pain (on the 100mm scale) compared to control group. 0 = no pain and 100 = worst pain imaginable.
Time Frame: Baseline, 3, 12, and 24 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Coflex™ | Surgical Decompression
Number analyzed (Participants) | 105 | 111
mm | -24.3 (2.5) | -20.6 (2.3)

5. Secondary Outcome: Neurological Status - Mean Change in Sensory Deficit From Baseline to 24 Months
Description: Sensory deficits will be assessed at nerves roots from L3, L4, L5, and S1. Grading score ranges from 1=absent to 3=normal.
Time Frame: Baseline, 3, 12, and 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coflex™ | Surgical Decompression
Number analyzed (Participants) | 105 | 111
score on a scale | 0.03 (0.01) | 0.04 (0.01)

6. Secondary Outcome: Assessment of Time to Symptoms Utilizing Walking Distance Test
Description: During this test, a patient has to walk on a treadmill (speed 1.8 km/h [12]) for 15 minutes (450 m) on a 0 degree ramp incline. It will be assessed time to first symptoms, time to severe symptoms and nature of symptoms (leg weakness, leg pain, back pain, or generalized fatigue, other). A time of zero will be recorded when symptoms were present at onset. The examination will be stopped after 15 minutes or at the onset of severe symptoms.
  Definition of severe symptoms is: The level of discomfort that would make patients stop their activities in usual life situations.
  It is assumed that patients with additional back pain will have more problems in managing the complete walking distance and therefore may stop the walking distance test before the endpoint at 15 minutes
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Coflex™ | Surgical Decompression
Number analyzed (Participants) | 105 | 111
minutes | 6.01 (0.65) | 4.36 (0.64)

7. Secondary Outcome: Number of Participants With Adverse Events - Operative Site
Description: Number of Participants that experience adverse events related to the operative site from each group.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Coflex™ | Surgical Decompression
Number analyzed (Participants) | 116 | 123
Participants | 45 | 54

8. Secondary Outcome: The Percentage of Patients With Survival Probability as Assessed by Evaluating Treatment Failure in Both Groups..
Description: Treatment failure is defined as any secondary intervention, severe adverse event or other parameters that define the device as ineffective or not safe. The following events/outcomes were defined as treatment failures: wound revisions, patients with trauma requiring surgical intervention, disc hernia or dura repair, and/or pain management.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Coflex™ | Surgical Decompression
Number analyzed (Participants) | 116 | 123
percentage of participants | 0.79 [0.70 to 0.85] | 0.76 [0.68 to 0.83]

9. Secondary Outcome: Change of Symptoms- Zurich Claudication Questionnaire (ZCQ) After 24 Months Compared to Baseline.
Description: The symptom severity scale ranges from 0 to 5 where a higher score indicates a worse outcome. Percentage of the maximum reported score for the symptom severity scale was calculated at baseline and 24 months and change in percentage score is reported in the Outcome Measure data table.
Time Frame: Baseline, 3, 12, and 24 months
Measure: Mean (Standard Deviation); unit: percentage points
Arm/Group | Coflex™ | Surgical Decompression
Number analyzed (Participants) | 105 | 111
percentage points | -15.0 (1.83) | -15.10 (1.75)

10. Secondary Outcome: Change in Functionality- Zurich Claudication Questionnaire (ZCQ) From Baseline to 24 Months
Description: as for outcome 9
Time Frame: Baseline, 3, 12, and 24 months
Measure: Mean (Standard Deviation); unit: percentage points
Arm/Group | Coflex™ | Surgical Decompression
Number analyzed (Participants) | 105 | 111
percentage points | -3.98 (0.38) | -3.52 (0.37)

11. Secondary Outcome: Neurological Status - Mean Change in Muscle Strength From Baseline to 24 Months
Description: Muscle strength will be assessed on right/left muscle strength at 6 groups of leg muscles. Score ranges from 0=contraction to 5=normal.
Time Frame: Baseline, Day 0 (Surgery), 3, 12, and 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coflex™ | Surgical Decompression
Number analyzed (Participants) | 105 | 111
score on a scale | 0.002 (0.035) | -0.030 (0.034)

12. Secondary Outcome: Assessment of Neurological Status Using the Laségue Test or Straight Leg Raise Test- Change From Baseline to 24 Months
Description: The straight leg raise or a Laségue Test is used to assess a participant's low back pain. A positive outcome is identified if a participant experiences low back pain when the straight leg is at a certain angle (0-90 degrees). A negative test suggests a likely different cause for back pain. The test is performed on both right and left legs.
Time Frame: Baseline, Day 0 (Surgery), 3, 12, and 24 months
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Coflex™ | Surgical Decompression
Number analyzed (Participants) | 105 | 111
Degrees | 10.8 (1.6) | 9.6 (1.6)

13. Secondary Outcome: Number of Participants Receiving Epidural Injections
Description: Epidural injections at up to 24 months
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Coflex™ | Surgical Decompression
Number analyzed (Participants) | 116 | 123
Participants | 0 | 2

14. Secondary Outcome: Neurological Status- Mean Change in Trendelenburg Sign Test From Baseline to 24 Months.
Description: Trendelenburg's sign was used to assess the neurological status of a subject. The test was taken for both the left and right sides and assessed as not present/absent (no= corresponding with a value of 1) or present (yes= corresponding to a value of 2). The average of each patient's worst side was calculated. Mean values closer to 1 indicate more patients with an absent Trendelenburg's sign, and a decrease in the mean change indicates more patients improving from a present to absent Trendelenburg's sign.
Time Frame: Baseline, Day 0 (Surgery), 3, 12, and 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coflex™ | Surgical Decompression
Number analyzed (Participants) | 105 | 111
score on a scale | -0.08 (0.36) | -0.05 (0.29)

15. Secondary Outcome: Neurological Status- Mean Change in Ilio Sacral Joint Affection Test From Baseline to 24 Months.
Description: Ilio sacral join affection test was used to assess the neurological status of a subject. The test was taken for both the left and right sides and assessed as not present/absent (no= corresponding with a value of 1) or present (yes= corresponding to a value of 2). The average of each patient's worst side was calculated. Mean values closer to 1 indicate more patients with an absent llio sacral joint affection and a decrease in the mean change indicates more patients improving from a present to absent sacral join affection.
Time Frame: Baseline, Day 0 (Surgery), 3, 12, and 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coflex™ | Surgical Decompression
Number analyzed (Participants) | 105 | 111
score on a scale | -0.10 (.43) | -0.07 (.45)

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse events were captured at either the operative site or non-operative site.
Arm/Group | Coflex™ | Surgical Decompression
All-Cause Mortality (participants affected / at risk) | 1/116 | 1/123
Serious Adverse Events (participants affected / at risk) | 89/116 | 96/123
Other Adverse Events (participants affected / at risk) | 89/116 | 96/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Coflex™ (N=116) | Surgical Decompression (N=123)
Gastritis (Gastrointestinal disorders) | 1 | 0 — Non-operative
Coxarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
Coronary Stent (Surgical and medical procedures) | 1 | 4 — Non-operative
APOPLECTIC STROKE ARTERIA CEREBRI MEDIA RIGHT (Nervous system disorders) | 2 | 0 — Non-operative
ARRYTHMIA ABSOLUTA (Cardiac disorders) | 1 | 0 — Non-operative
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — Non-operative
CARDIAC ARRHYTHMIA (Cardiac disorders) | 1 | 0 — Non-operative
CARDIAC STENT (Cardiac disorders) | 1 | 0 — Non-operative
CATARACT LEFT EYE (Eye disorders) | 1 | 0 — Non-operative
CERVICAL DISC HERNIATION (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
COLITIS (Gastrointestinal disorders) | 1 | 1 — Non-operative
STOMACH POLYP (Gastrointestinal disorders) | 1 | 0 — Non-operative
FACET PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
FALL (Injury, poisoning and procedural complications) | 1 | 0 — Non-operative
FRACTURE PROXIMAL HUMERUS SURGERY (PLATE) (Surgical and medical procedures) | 1 | 0 — Non-operative
FUSION C5/C6 (Surgical and medical procedures) | 1 | 0 — Non-operative
GENERAL WEAKNESS (General disorders) | 1 | 0 — Non-operative
HEART ATTACK (Cardiac disorders) | 1 | 0 — Non-operative
HIP ARTHROSIS LEFT (Musculoskeletal and connective tissue disorders) | 2 | 0 — Non-operative
HIP SURGERY, KNOWN COXARTHROSIS (Surgical and medical procedures) | 1 | 0 — Non-operative
IMPLANTATION CORONARY STENT (Surgical and medical procedures) | 1 | 0 — Non-operative
IMPLANTATION OF TEP LEFT HIP (Surgical and medical procedures) | 1 | 0 — Non-operative
KNEE PAIN AND SURGERY LEFT 08 JUN 2011 (Surgical and medical procedures) | 1 | 0 — Non-operative
LEG PAIN RIGHT (GLUTEAL PAIN RIGHT SIDE) (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
LENS EXCHANGE RIGHT EYE (Surgical and medical procedures) | 1 | 0 — Non-operative
LUMBAR BACK PAIN L5/S1 AND L3/L4 (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
MILD HEAD INJURY (Injury, poisoning and procedural complications) | 1 | 0 — Non-operative
MYASTHENIA GRAVIS (Nervous system disorders) | 1 | 0 — Non-operative
MYELODYSPLASIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — Non-operative
MYELOPATHY CERVICULAR WITH SPONDYLODESIS C3/4 (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 0 — Non-operative
NASAL SEPTUM DEVIATION (Injury, poisoning and procedural complications) | 1 | 0 — Non-operative
NEPHROLITHIASIS LEFT (Renal and urinary disorders) | 1 | 0 — Non-operative
PACE-MAKER-IMPLANTATION (Surgical and medical procedures) | 1 | 0 — Non-operative
PATIENT FELL DOWN, CONTUSION OF RIGHT FEMUR AND HIP (Injury, poisoning and procedural complications) | 1 | 0 — Non-operative
PERIPHERAL ARTERIAL DISEASE BOTH LEGS (Vascular disorders) | 1 | 0 — Non-operative
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Non-operative
PNEUMONIA WITH RENAL FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Non-operative
PSYCHOTIC SYNDROME (Psychiatric disorders) | 1 | 0 — Non-operative
PUPIL INFARCTION (Eye disorders) | 1 | 0 — Non-operative
RADIUSFRACTURE LEFT (Injury, poisoning and procedural complications) | 1 | 0 — Non-operative
RESECTION OF NOSE POLYPOSIS (Surgical and medical procedures) | 1 | 0 — Non-operative
RIB FRACTURE WITH PNEUMONIA (Infections and infestations) | 1 | 0 — Non-operative
S1 Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
SECOND REVISION OF THE KNEE-TEP RIGHT SIDE (Surgical and medical procedures) | 1 | 0 — Non-operative
STENOSIS ARTERIA FEMORALIS / PERIPHERAL ARTERIAL VENOUS DISEASE (Vascular disorders) | 1 | 0 — Non-operative
STENOSIS DUCTUS HEPATOCHOLEDOCHUS (Hepatobiliary disorders) | 1 | 0 — Non-operative
STENTS AND DILATATION (Surgical and medical procedures) | 1 | 0 — Non-operative
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 1 | 0 — Non-operative
SYNCOPE (Cardiac disorders) | 1 | 0 — Non-operative
TOTAL RESECTION UTERUS (Surgical and medical procedures) | 1 | 0 — Non-operative
TRANSIENT ISCHEMIC ATTACK (Cardiac disorders) | 1 | 0 — Non-operative
VASCULAR STENOSIS (VASCULAR STENT INGUINAL LEFT) (Surgical and medical procedures) | 1 | 0 — Non-operative
COMPONENT MIGRATION (Injury, poisoning and procedural complications) | 1 | 0 — Operative
DISC HERNIATION L5/S1 LEFT (Musculoskeletal and connective tissue disorders) | 1 | 0 — Operative
DISC HERNIATION SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 — Operative
DURAL VIOLATION (Injury, poisoning and procedural complications) | 1 | 1 — Operative
FRACTURE PROC SPINOSUS (Injury, poisoning and procedural complications) | 1 | 0 — Operative
FRACTURE, SPECIFY: FRACTURE SPINOUS PROCESS (Injury, poisoning and procedural complications) | 1 | 0 — Operative
FRACTURE, SPECIFY: SPINOUS PROCESS FRACTURE L4 (Injury, poisoning and procedural complications) | 1 | 0 — Operative
HEMATOMA REQUIRING DRAINAGE (Blood and lymphatic system disorders) | 2 | 1 — Operative
INFECTION (DEEP) DEEP WOUND INFECTION (Infections and infestations) | 1 | 0 — Operative
NERVE INJURY (Injury, poisoning and procedural complications) | 1 | 0 — Operative
DEGENERATION NEIGHBORING SEGMENTS (Musculoskeletal and connective tissue disorders) | 1 | 0 — Operative
INCREASE BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 — Operative
LUMBAR PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 — Operative
RECURRENT PAIN (General disorders) | 1 | 0 — Operative
SPONDYLODICITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 — Operative
SUPERFICIAL WOUND INFECTION (Infections and infestations) | 1 | 0 — Operative
SYNOVIAL CYSTS (Musculoskeletal and connective tissue disorders) | 2 | 0 — Operative
BACK PAIN DUE TO ILIOSACRAL JOINT AFFECTION (Musculoskeletal and connective tissue disorders) | 1 | 0 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BACK LUMBAR PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BACK PAIN CONTINUED WITH FUSION L3-S1 (Musculoskeletal and connective tissue disorders) | 1 | 0 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BOTH LEG AND BACK LEG AND BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BOTH LEG AND BACK LEG PAIN LEFT AND RIGHT, BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 — Operative
TRAUMA FRACTURE L2, NUCLEUS-PULPOSUS-PROLAPS L4/5 LEFT (Musculoskeletal and connective tissue disorders) | 1 | 0 — Operative
L1 FRACTURE AFTER TRAUMA (Injury, poisoning and procedural complications) | 1 | 0 — Operative
WOUND PROBLEMS (Infections and infestations) | 3 | 3 — Operative
CATARACT (EYE SURGERY) (Surgical and medical procedures) | 1 | 0 — Non-operative
ENDOSCOPIC SURGERY STOMACH POLYP (Surgical and medical procedures) | 1 | 0 — Non-operative
INFECTION (DEEP) (Infections and infestations) | 2 | 1 — Operative
WOUND PROBLEMS PROLONGED SECRETOR (Infections and infestations) | 1 | 0 — Operative
CORONARY HEART DISEASE - BYPASS SURGERY (Surgical and medical procedures) | 0 | 1 — Non-operative
ARRHYTHMIA (Cardiac disorders) | 0 | 1 — Non-operative
ILIOSACRAL JOINT AFFECTION LEFT WITH NEED FOR DENERVATION (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
KNEE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
PULMONARY EMBOLISM (Cardiac disorders) | 0 | 1 — Non-operative
ARRHYTHMIA (PACEMAKER IMPLANTATION) (Surgical and medical procedures) | 0 | 1 — Non-operative
LITTLE APOPLEXY (Cardiac disorders) | 0 | 1 — Non-operative
PROSTATA CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — Non-operative
PAIN TESTICLE (ORCHIECTOMY LEFT) (Surgical and medical procedures) | 0 | 1 — Non-operative
ALCOHOL WITHDRAWAL DELIRIUM AURICULAR FIBRILLATION (Psychiatric disorders) | 0 | 1 — Non-operative
DYSPNOE BECAUSE OF ASTHMA (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
HIP PROSTHESIS LEFT, COXARTHROSIS LEFT (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
REPLACEMENT OF RIGHT HIP PROSTHESIS, DYSFUNCTION OF HIP PROSTHESIS (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
OPERATION RIGHT SHOULDER (Surgical and medical procedures) | 0 | 1 — Non-operative
KNEE OPERATION LEFT (Surgical and medical procedures) | 0 | 1 — Non-operative
KNEE PROSTHESIS LEFT (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
NEW OCCURRENCE OF ISCHIALGIA LEFT LEG WITH HYPAESTHESIA LEFT LEG (Nervous system disorders) | 0 | 1 — Non-operative
PAIN OF LEFT HIP, ENDOPROSTHESIS (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
HYPAESTHESIA (WITH ACUTE PAIN LEFT LEG) (Nervous system disorders) | 0 | 1 — Non-operative
NEUROLOGIC DISORDER (Nervous system disorders) | 0 | 1 — Non-operative
FRACTURE THORACIC VERTEBRA NO.12 (Injury, poisoning and procedural complications) | 0 | 1 — Non-operative
PAINFUL LEG WITH ELECTIVE ANGIOGRAPHY, FEMORAL ARTERIAL STENOSIS (Vascular disorders) | 0 | 1 — Non-operative
GASTRIC BLEEDING (Gastrointestinal disorders) | 0 | 1 — Non-operative
COXARTHROSIS, HIP TOTAL ENDOPROTHESIS (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
VIRUS PNEUMONIA (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
TUBERCULOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
HYPERTENSIVE CRISIS (Cardiac disorders) | 0 | 1 — Non-operative
KNEE PAIN, TOTAL ENDOPROSTHESIS LEFT PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
HYPERTONUS (Cardiac disorders) | 0 | 1 — Non-operative
HOSPITALIZATION DUE TO PARESIS (Nervous system disorders) | 0 | 1 — Non-operative
UROLOGIC PROBLEMS (PROSTATIC HYPERPLASIA) (Renal and urinary disorders) | 0 | 1 — Non-operative
GONARTHROSIS (TEP LEFT KNEE) (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
COLON INFECTION (Gastrointestinal disorders) | 0 | 1 — Non-operative
2 STENTS (Cardiac disorders) | 0 | 1 — Non-operative
CHOLECYSTITIS (Renal and urinary disorders) | 0 | 1 — Non-operative
ENDOSCOPIC EXPLORATION FOR LYMPHATIC NOTCH HISTOLOGY (Surgical and medical procedures) | 0 | 1 — Non-operative
TOTAL ENDOPROSTHESIS RIGHT HIP (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
GONALGIA LEFT (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
KNOWN COXARTHROSIS WITH TEP (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
APOPLEXY (Nervous system disorders) | 0 | 2 — Non-operative
CHRONICAL MYELOMA PROLIFERATIVE DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — Non-operative
RELAPSE OF RECTUM CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — Non-operative
PAIN AND SWELLING LEFT ANKLE (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
PROGRESSION OF GONARTHROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
PANCREAS TUMOR AND PANCREAS SURGERY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — Non-operative
GONARTHROSIS, KNEE PROSTHESIS LEFT 01. JUNE 2011 (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
KNEE ARTHROSIS RIGHT (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
PEMPHIGUS, BASALIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — Non-operative
HIP INJURY (Injury, poisoning and procedural complications) | 0 | 1 — Non-operative
CANCER ESOPHAGUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — Non-operative
CATARACT (Eye disorders) | 0 | 1 — Non-operative
HIP PROSTHESIS (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
RADIUS FRACTURE RIGHT (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
HERPES ZOSTER (Infections and infestations) | 0 | 1 — Non-operative
AORTIC ANEURYSM (Cardiac disorders) | 0 | 1 — Non-operative
LUMBAR PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BACK LUMBAR PAIN ILIOSACRAL JOINT AFFECTION (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BOTH LEG AND BACK FACET DENERVATION L2-S1 (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
DISC HERNIATION DISC HERNIATION (Musculoskeletal and connective tissue disorders) | 0 | 3 — Operative
SPONDYLODESIS L4/L5 AUGUST 2015 (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BOTH LEG AND BACK PERSISTENT BACK AND LEG PAIN L2-5 (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - LEG LEG PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BOTH LEG AND BACK INCREASE PAIN BACK, LEGS (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BACK ACUTE INCREASE OF PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BACK CONTINUOUS DEGENERATION OF LUMBAL SPINE (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
DISC HERNIATION HERNIATED VERTEBRAL DISC (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
RESTENOSIS (Blood and lymphatic system disorders) | 0 | 1 — Operative
CEREBROSPINAL FLUID CYST (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - LEG ISCHIALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BACK BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BACK RADICULOPATHY AND INCREASING BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
INCREASING VENTROLISTHESIS L4/5 (Musculoskeletal and connective tissue disorders) | 0 | 2 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BOTHAEMATOMA WITH LUMBAGO AND ISCHIALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - LEG COMPRESSION (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BOTH LEG AND BACK LUMBAGO ISCHIALGIA LEFT (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BOTH LEG AND BACK DEGENERATION L4-S1 (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BACK PAIN, INSTABILITY (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BOTH LEG AND BACK INCREASING LEG AND BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
TRAUMA FALL WITH LUMBAR FRACTURES (Injury, poisoning and procedural complications) | 0 | 1 — Operative
BACK PAIN, LEFT LEG PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Coflex™ (N=116) | Surgical Decompression (N=123)
TRAUMA FALL (Injury, poisoning and procedural complications) | 1 | 0 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BOTH LEG AND BACK BACK PAIN, POSSIBLE BECAUSE OF KNEE PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Operative
CEREBROSPINAL FLUID LEAKAGE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Operative
LOCAL OSTEOPOROSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BACK INCREASING BACK PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Operative
DISC HERNIATION DISC PROLAPS L4/5 (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Operative
TRAUMA BACK PAIN AFTER FALL (Injury, poisoning and procedural complications) | 1 | 0 — Operative
SACROILIAC JOINT PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Operative
WOUND PROBLEMS (Infections and infestations) | 6 | 5 — Operative
DURAL VIOLATION (Injury, poisoning and procedural complications) | 3 | 19 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BACK INCREASING LUMBAGO (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BOTH LEG AND BACK LUMBOISCHIALGIA LEFT (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Operative
COMPONENT MIGRATION DORSAL MIGRATION OF COFLEX (Injury, poisoning and procedural complications) | 1 | 0 — Operative
FRACTURE, SPECIFY: TIIP OF SPINOUS PROCESS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Operative
PROGRESSIVE OSTEOCHONDROSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Operative
FRACTURE, SPECIFY: FISSURE (Injury, poisoning and procedural complications) | 1 | 0 — Operative
DURAL VIOLATION L5/S1 (Injury, poisoning and procedural complications) | 1 | 0 — Operative
COXALGIA LEFT (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
VERTIGO (Nervous system disorders) | 1 | 0 — Non-operative
FALL WITH FOLLOWING BACK PAIN (Injury, poisoning and procedural complications) | 1 | 0 — Non-operative
TROCHANTER PAIN BOTH SIDES RESP. PELVIC + HIP PAIN BOTH SIDES (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
HIP PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 — Non-operative
KNEE PAIN BOTH SIDES (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
PAIN KNEE (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
RENAL INSUFFICIENCY (Renal and urinary disorders) | 1 | 0 — Non-operative
INFECTION INTESTINAL WITH CLOSTRIDIA (Gastrointestinal disorders) | 1 | 0 — Non-operative
GONARTHROSIS BOTH (Musculoskeletal and connective tissue disorders) | 2 | 0 — Non-operative
DISORIENTATION CEREBRAL (Nervous system disorders) | 1 | 0 — Non-operative
PAIN RIGHT HIP (Musculoskeletal and connective tissue disorders) | 3 | 1 — Non-operative
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1 — Non-operative
BLADDER DYSFUNCTION (Renal and urinary disorders) | 1 | 0 — Non-operative
EDEMA LOWER LEGS (Blood and lymphatic system disorders) | 1 | 0 — Non-operative
ANGINA PECTORIS (Cardiac disorders) | 1 | 0 — Non-operative
GONARTHROSIS ACTIVATED (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
CORPUS VITREUM RETRACTION (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
CRAMPS IN THIGHS (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
SYMPTOMATIC TRANSITORY PSYCHOTIC SYNDROME (Psychiatric disorders) | 1 | 0 — Non-operative
DIZZINESS (General disorders) | 1 | 0 — Non-operative
DIABETES MELLITUS (Endocrine disorders) | 1 | 0 — Non-operative
MUSCLE INJURY LEFT GLUTEAL (Injury, poisoning and procedural complications) | 1 | 0 — Non-operative
ALLERGIC EXANTHEMA (Endocrine disorders) | 1 | 0 — Non-operative
GONARTHROSIS LEFT (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
PERIPHERAL ARTERIAL DISEASE (Cardiac disorders) | 1 | 0 — Non-operative
BAD VIEW DUE TO DIABETES (Endocrine disorders) | 1 | 0 — Non-operative
BYPASS LEG DUE TO PERIPHERAL ARTERIAL DISEASE (Surgical and medical procedures) | 1 | 0 — Non-operative
FRACTURE OF LEFT HAND, OS TRIQUETRUM AVULSION FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
HIP PAIN AFTER TOTAL HIP REPLACEMENT 2003 (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
DISCS HERNIATION CERVICAL VERTEBRAL BODY 6/7 (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Non-operative
FALL (Injury, poisoning and procedural complications) | 1 | 0 — Non-operative
COXARTHROSIS LEFT (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
HERPES LABIALIS (Infections and infestations) | 1 | 0 — Non-operative
CARDIAC INSUFFICIENCY (Cardiac disorders) | 1 | 0 — Non-operative
CARPAL TUNNEL SYNDROME RIGHT (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
CERVICAL MYELOPATHY (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — Non-operative
ILIO-SACRAL JOINT AFFECTION (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
PAIN BURSA TROCHANTERICA RIGHT (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
BURSITIS TROCHANTERICA LEFT (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Non-operative
POLYNEUROPATHY (Nervous system disorders) | 1 | 2 — Non-operative
INCREASING COXARTHROSIS RIGHT (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
SCAPHOID-TRAPEZIUM-ARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
SCLEROSIS OF HAEMORRHOIDS (Skin and subcutaneous tissue disorders) | 1 | 0 — Non-operative
HYPERTENSION (Cardiac disorders) | 2 | 0 — Non-operative
ANEMIA (Cardiac disorders) | 1 | 0 — Non-operative
PAIN LEFT KNEE (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
KNEE PAIN AFTER FALL (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
BREACKAGE OF A RIP (Investigations) | 1 | 0 — Non-operative
FRACTURE RIGHT HAND (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
KNEE ARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
PSYCHOSYNDROME (Psychiatric disorders) | 1 | 0 — Non-operative
POOR GENERAL HEALTH STATUS (General disorders) | 1 | 0 — Non-operative
FINGER ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
URINARY INFECTION (Infections and infestations) | 1 | 1 — Non-operative
KNEE PAIN LEFT (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
PAIN RIGHT KNEE (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
CRAMP PAIN AND DYSESTHESIA IN BOTH FEET (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
HIP ARTHROSIS LEFT (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 — Non-operative
GASTROINTESTINAL INFECT (Gastrointestinal disorders) | 1 | 0 — Non-operative
POTENTIAL HIP ARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
LEG PAIN LEFT >> RIGHT (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
UNKNOWN SYNCOPE (Cardiac disorders) | 1 | 0 — Non-operative
ACUTE HEARING LOSS (Ear and labyrinth disorders) | 1 | 0 — Non-operative
MENISCUS OPERATION RIGHT - CAUSE OF KNEE PAIN (Surgical and medical procedures) | 1 | 0 — Non-operative
MILD PAIN LEFT THIGH (Musculoskeletal and connective tissue disorders) | 1 | 0 — Non-operative
BLADDER DISTURBANCE (Renal and urinary disorders) | 1 | 0 — Non-operative
BURSITIS TROCHANTERICA RIGHT (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Non-operative
FEELING OF WEAKNESS IN BOTH KNEES (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
HIP PAIN INCREASING (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
DEPRESSION INTERMITTENT (Psychiatric disorders) | 0 | 1 — Non-operative
FACET INFILTRATION L3/4 + L5/S1 (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
ACUTE PAIN LEFT LEG (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
CRISIS OF HYPERTENSION (Cardiac disorders) | 0 | 1 — Non-operative
PAINFUL RIGHT LEG (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
OMARTHROSIS LEFT (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
CERVICAL SYNDROME WITH MIGRAINE (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
PSEUDORADIKULARSYNDROM (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
CERVICAL SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
HYSTERIC PTOSIS (Reproductive system and breast disorders) | 0 | 1 — Non-operative
HYPERTENSIVE CRISIS (Cardiac disorders) | 0 | 1 — Non-operative
PARALYSIS DIAPHRAGM LEFT (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Non-operative
HIP PAIN LEFT (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
PARASTHESIA FOREFOOT BOTH SIDES (Nervous system disorders) | 0 | 1 — Non-operative
HAGLUND HEEL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
ANEMIA (Blood and lymphatic system disorders) | 0 | 1 — Non-operative
NERVOUS BREAK DOWN (Psychiatric disorders) | 0 | 1 — Non-operative
PARESTHESIA FOREFOOT RIGHT (Nervous system disorders) | 0 | 1 — Non-operative
ARTERIAL STENOSIS LEFT POPLITEA (Vascular disorders) | 0 | 1 — Non-operative
GONARTHROSIS (Musculoskeletal and connective tissue disorders) | 0 | 2 — Non-operative
CERATOACANTHOMA SURGERY (Surgical and medical procedures) | 0 | 1 — Non-operative
PSYCHOSIS, ALCOHOL ABUSE (Psychiatric disorders) | 0 | 1 — Non-operative
SUSPECT OF SEIZURES (Nervous system disorders) | 0 | 1 — Non-operative
FOOT PAIN ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
BLADDER INFECTION/URINARY TRACT INFECTION (Renal and urinary disorders) | 0 | 1 — Non-operative
HIP AND KNEE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
COXARTHROSIS (Musculoskeletal and connective tissue disorders) | 0 | 2 — Non-operative
BASALIOMA SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — Non-operative
GLAUCOMA BOTH SIDES (Eye disorders) | 0 | 1 — Non-operative
PAIN RIGHT EAR (Ear and labyrinth disorders) | 0 | 1 — Non-operative
HYPERTENSION (Cardiac disorders) | 0 | 1 — Non-operative
ALLERGIC REACTION TO PLASTER (Endocrine disorders) | 0 | 1 — Non-operative
PAIN IN NECK (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
VERTIGO (Nervous system disorders) | 0 | 2 — Non-operative
CHEST-PAIN (Cardiac disorders) | 0 | 1 — Non-operative
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Non-operative
PROGRESSIVE ARTERIAL DISSEASE (Vascular disorders) | 0 | 1 — Non-operative
CRAMPS IN LEGS (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
ONYCHECTOMY DIGIT 2 RIGHT HAND (Surgical and medical procedures) | 0 | 1 — Non-operative
HAEMANGIOMA LEFT EYE (Eye disorders) | 0 | 1 — Non-operative
ANKLE SPRAIN LEFT (Injury, poisoning and procedural complications) | 0 | 1 — Non-operative
DEPRESSION (Psychiatric disorders) | 0 | 1 — Non-operative
CEPHALGIA WITH CERVICOBRACHIALGIA, SYNDROME (Nervous system disorders) | 0 | 1 — Non-operative
BASALIOM LEFT EAR (Ear and labyrinth disorders) | 0 | 1 — Non-operative
TRICEPS TENDON RUPTURE (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
COXARTHROSIS RIGHT WITH HIP PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
ORTHOSTATIC DYSREGULATION (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
L2 OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
ARTHRITIS LEFT KNEE (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
CERVICOBRACHIAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
DIZZINESS (General disorders) | 0 | 1 — Non-operative
PAIN IN BOTH KNEES AFTER FALL (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
LIVER CANCER, KNOWN CIRRHOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — Non-operative
KNEE PAIN LEFT (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-operative
DIAGNOSIS OF ENCEPHALOPATHY (MULTIPLE SCLEROSIS) (Nervous system disorders) | 0 | 1 — Non-operative
BRACHIALGIA RIGHT (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Non-operative
BRACHIALGIA LEFT ARM (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Non-operative
KNEE PAIN RIGHT (Respiratory, thoracic and mediastinal disorders) | 0 | 2 — Non-operative
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Non-operative
CAR ACCIDENT WITH CERVICAL PAIN (Injury, poisoning and procedural complications) | 0 | 1 — Non-operative
PAIN; NEW, AND FREQUENCY, WORSENING - BACK LUMBAGO, FACET-SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
DISCUS PROTRUSION L5/6 (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
NEVE INJURY PARAESTHESIA LEGS (Nervous system disorders) | 0 | 1 — Operative
HEMATOMA REQUIRING DRAINAGE (Blood and lymphatic system disorders) | 0 | 1 — Operative
CYST OF FACET JOINT (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - LEG LEG PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
HETROTOPIC OSSIFICATION (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
WOUND PROBLEMS BULKY SCAR (Infections and infestations) | 0 | 1 — Operative
DURAL VIOLATION SMALL LEAK OF DURA INTEROPERATIVE L3/4 (Injury, poisoning and procedural complications) | 0 | 1 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BACK ILIO SACRAL JOINT AFFECTION BOTH SIDES (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
PAIN; NEW, AND FREQUENCY, WORSENING - BACK LUMBAGO (Musculoskeletal and connective tissue disorders) | 0 | 1 — Operative
INCREASING ISCHIALGIA (Nervous system disorders) | 0 | 1 — Operative
NERVE AFFECTION (Nervous system disorders) | 0 | 1 — Operative

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No